CLINICAL TRIAL: NCT00855959
Title: An Evaluation of Efficacy and Safety of Corresponding Doses of Pulmicort Turbuhaler® and Pulmicort Respules® in Japanese Asthmatic Adult Patients (Open, Multicenter, Phase III Study)
Brief Title: Study to Evaluate Efficacy and Safety of Pulmicort Respules in Japanese Adult Asthmatic Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Carlsson, Lars-Goran, MD, Medical Science Director, Est.Respiratory Brands, AstraZeneca Pharmaceuticals
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D5259C00001
Record Dates: First submitted 2009-03-04; First posted 2009-03-05 (Estimated); Results first posted 2011-03-11 (Estimated); Last update posted 2011-03-11 (Estimated); Status verified 2011-02

CONDITIONS: Asthma
Keywords: Asthma; Pulmicort Respules
MeSH Terms: conditions — Asthma | interventions — Budesonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Four weeks treatment with either Pulmicort Turbuhaler at a dose of 400 μg or 200 ug twice daily, followed by 6 weeks treatment with Pulmicort Respules at a dose of 1.0 mg twice daily or 0.5 mg twice daily/1.0 mg once daily
  Interventions: Drug: Budesonide
- 2 (Experimental): Pulmicort Turbuhaler at a dose of 200 μg twice daily and Pulmicort Respules at a dose of 0.5 mg twice daily or 1.0 mg once daily (low dose)
  Interventions: Drug: Pulmicort Turbuhaler

INTERVENTIONS:
Drug: Budesonide — Inhalation powder, inhalation, twice daily, 4 weeks followed by Suspension for nebulisation, inhalation, once or twice daily, 6 weeks
  Other Names: Pulmicort
  Arms: 1
Drug: Pulmicort Turbuhaler — Pulmicort Turbuhaler 200 µg, Dry powder inhaler, budesonide 200 µg/dose, 112 doses/Turbuhaler
  Arms: 2

SUMMARY:
The primary objective of the study is to show similarity of efficacy on Pulmicort Respules 1.0 mg/day or 2.0 mg/day for 6 weeks in the treatment period and the corresponding doses of Pulmicort Turbuhaler 400 μg/day or 800 μg/day for 4 weeks in the observation period in Japanese adult asthmatic patients with age of 16 years or older.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent prior to any study specific procedures.
* A minimum of 6 months documented history of asthma according to the JGL 2006 definition
* Asthma patients under prescribed treatment with ICS at least 3 months before Visit 2.

Exclusion Criteria:

* Current or previous tobacco smokers with a history of >= 10 pack-years
* Use of β-blockers including eye drops
* Clinically significant respiratory infection affecting the asthma, as judged by the investigator(s) within 4 weeks prior to visit 2
* Intake of oral, rectal or parenteral GCS within 4 weeks prior to Visit 2

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2009-02; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lars-Göran Carlsson, MD, Study Director — AstraZeneca R&D Lund
Locations (6):
- Japan (6):
  - Research Site, Ichikawa, Chiba
  - Research Site, Yokosuka, Kanagawa
  - Research Site, Chiyoda City, Tokyo
  - Research City, Hino, Tokyo
  - Research Site, Setagaya City, Tokyo
  - Research Site, Tachikawa, Tokyo

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Outpatients, male and female ≥ 16 years with stable asthma
Groups:
- Pulmicort Turbuhaler and Pulmicort Respules: 4 weeks treatment with either Pulmicort Turbuhaler at a dose of 400 μg or 200 ug twice daily, followed by 6 weeks treatment with Pulmicort Respules at a dose of 1.0 mg twice daily or 0.5 mg twice daily/1.0 mg once daily
Period: Overall Study
Arm/Group | Pulmicort Turbuhaler and Pulmicort Respules
Started | 108
Patients Who Received Pulmicort Respules | 105
Completed | 99
Not Completed | 9
Not completed — Adverse Event | 2
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 3
Not completed — Pregnancy | 1
Not completed — Incorrect enrolment | 1

BASELINE CHARACTERISTICS:
Arm/Group | Pulmicort Turbuhaler and Pulmicort Respules
Number analyzed (Participants) | 106
Age Continuous [Mean (Standard Deviation); unit: Years] | 43.9 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73
  Male | 33

OUTCOME MEASURES:

1. Primary Outcome: Morning Peak Expiratory Flow (mPEF)
Description: Change in morning peak expiratory flow (mPEF) from baseline (mean of the last 14 days of the period on Pulmicort Turbuhaler) to Week 6 (mean of the last 14 days of the period on Pulmicort Respules)
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | Pulmicort Turbuhaler and Pulmicort Respules
Number analyzed (Participants) | 105
L/min | 3.3 (21.4)

2. Secondary Outcome: Evening Peak Expiratory Flow (ePEF)
Description: Change in evening peak expiratory flow (ePEF) from baseline (mean of the last 14 days of the period on Pulmicort Turbuhaler) to Week 6 (mean of the last 14 days of the period on Pulmicort Respules)
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | Pulmicort Turbuhaler and Pulmicort Respules
Number analyzed (Participants) | 105
L/min | 3.8 (18.1)

3. Secondary Outcome: Asthma Symptom Score (Daytime); Score of 0-3 (0 = no Asthma Symptoms - 3 = Severe Symptoms)
Description: Change in Asthma symptom score (Daytime) from baseline (mean of the last 14 days of the period on Pulmicort Turbuhaler) to Week 6 (mean of the last 14 days of the period on Pulmicort Respules)
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Pulmicort Turbuhaler and Pulmicort Respules
Number analyzed (Participants) | 105
Scores on a scale | 0.018 (0.198)

4. Secondary Outcome: Asthma Symptom Score (Night-time); Score of 0-3 (0 = no Asthma Symptoms - 3 = Severe Symptoms)
Description: Change in Asthma symptom score (Night-time) from baseline (mean of the last 14 days of the period on Pulmicort Turbuhaler) to Week 6 (mean of the last 14 days of the period on Pulmicort Respules)
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Pulmicort Turbuhaler and Pulmicort Respules
Number analyzed (Participants) | 105
Scores on a scale | 0.022 (0.185)

5. Secondary Outcome: Asthma Symptom Score (Total); Score of 0-3 (0 = no Asthma Symptoms - 3 = Severe Symptoms)
Description: Change in Asthma symptom score (Total) from baseline (mean of the last 14 days of the period on Pulmicort Turbuhaler) to Week 6 (mean of the last 14 days of the period on Pulmicort Respules)
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Pulmicort Turbuhaler and Pulmicort Respules
Number analyzed (Participants) | 105
Scores on a scale | 0.039 (0.346)

6. Secondary Outcome: Use of Rescue Medication (Daytime)
Description: Change in Use of rescue medication (Daytime) from baseline (mean of the last 14 days of the period on Pulmicort Turbuhaler) to Week 6 (mean of the last 14 days of the period on Pulmicort Respules)
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: puffs
Arm/Group | Pulmicort Turbuhaler and Pulmicort Respules
Number analyzed (Participants) | 105
puffs | 0.017 (0.160)

7. Secondary Outcome: Use of Rescue Medication (Night-time)
Description: Change in Use of rescue medication (Night-time) from baseline (mean of the last 14 days of the period on Pulmicort Turbuhaler) to Week 6 (mean of the last 14 days of the period on Pulmicort Respules)
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: puffs
Arm/Group | Pulmicort Turbuhaler and Pulmicort Respules
Number analyzed (Participants) | 105
puffs | 0.044 (0.220)

8. Secondary Outcome: Use of Rescue Medication (Total)
Description: Change in Use of rescue medication (Total) from baseline (mean of the last 14 days of the period on Pulmicort Turbuhaler) to Week 6 (mean of the last 14 days of the period on Pulmicort Respules)
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: puffs
Arm/Group | Pulmicort Turbuhaler and Pulmicort Respules
Number analyzed (Participants) | 105
puffs | 0.061 (0.317)

9. Secondary Outcome: Night-time Awakenings Due to Asthma Symptoms
Description: Change in Night-time awakenings due to asthma symptoms from baseline (mean of the last 14 days of the period on Pulmicort Turbuhaler) to Week 6 (mean of the last 14 days of the period on Pulmicort Respules)
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: awakenings
Arm/Group | Pulmicort Turbuhaler and Pulmicort Respules
Number analyzed (Participants) | 105
awakenings | -0.004 (0.165)

10. Secondary Outcome: Forced Expiratory Volume in 1 Second (FEV 1.0)
Description: Change in Forced Expiratory Volume in 1 second (FEV 1.0) from baseline (mean of the last 14 days of the period on Pulmicort Turbuhaler) to Week 6 (mean of the last 14 days of the period on Pulmicort Respules)
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Pulmicort Turbuhaler and Pulmicort Respules
Number analyzed (Participants) | 102
L | 0.079 (0.244)

11. Secondary Outcome: Forced Vital Capacity (FVC)
Description: Change in Forced Vital Capacity (FVC) from baseline (mean of the last 14 days of the period on Pulmicort Turbuhaler) to Week 6 (mean of the last 14 days of the period on Pulmicort Respules)
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Pulmicort Turbuhaler and Pulmicort Respules
Number analyzed (Participants) | 102
L | 0.105 (0.283)

12. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: Number of participants with AEs reported during the period on Pulmicort Respules
Time Frame: 6 weeks
Measure: Number; unit: Participants
Arm/Group | Pulmicort Turbuhaler and Pulmicort Respules
Number analyzed (Participants) | 105
Participants | 50

ADVERSE EVENTS:
Arm/Group | Pulmicort Turbuhaler and Pulmicort Respules
Serious Adverse Events (participants affected / at risk) | 0/108
Other Adverse Events (participants affected / at risk) | 7/105
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pulmicort Turbuhaler and Pulmicort Respules (N=105)
Nasopharyngitis (Renal and urinary disorders) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less